CLINICAL TRIAL: NCT06918912
Title: Use of LOncastuximab Tesirine in Patients With RElapsed/Refractory Diffuse LargeB-Cell LYmphoma (DLBCL) or High Grade B-Cell Lymphoma (HGBCL) Who Have Progressive Disease After CAR T-cell Treatment
Brief Title: Study of Loncastuximab Tesirine in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) or High-Grade B-Cell Lymphoma (HGBCL) Following CAR-T Therapy Failure
Acronym: LORELY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2021-001; 2024-516929-31-00 (EU CTIS Number); 2022-001147-24 (EudraCT Number)
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B-Cell Lymphoma; High-grade B-cell Lymphoma (HGBCL); B-Cell Lymphoma Treatment; Relapsed or Refractory Lymphoma
Keywords: Antibody-Drug Conjugates; Loncastuximab Tesirine
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Loncastuximab Tesirine in Relapsed/Refractory DLBCL or HGBCL after CAR-T Failure (Experimental): This arm of the study involves the administration of Loncastuximab Tesirine to patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) or High-Grade B-Cell Lymphoma (HGBCL) who have failed prior treatment with CAR-T therapy. Participants will receive an intravenous infusion of Loncastuximab Tesirine at a dose of 150 μg/kg for the first two cycles, followed by 75 μg/kg for up to 6 additional cycles, totaling 8 cycles of treatment. The drug will be administered every 3 weeks. The primary goal is to evaluate the treatment's efficacy, as well as its safety, by monitoring response rates, progression-free survival, and overall survival, along with potential adverse events. Participants will be followed for 24 months after the end of treatment.
  Interventions: Drug: Loncastuximab Tesirine (Anti-CD19 Antibody-Drug Conjugate)

INTERVENTIONS:
Drug: Loncastuximab Tesirine (Anti-CD19 Antibody-Drug Conjugate) — Loncastuximab Tesirine is an antibody-drug conjugate specifically targeting CD19, a protein found on the surface of B-cells. It is designed to deliver a cytotoxic pyrrolobenzodiazepine dimer directly to CD19-expressing malignant B-cells. Unlike traditional chemotherapies, Loncastuximab Tesirine combines the precision of an anti-CD19 monoclonal antibody with a potent chemotherapy agent, offering targeted therapy for relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) and High-Grade B-Cell Lymphoma (HGBCL) after failure of CAR-T therapy. It is administered intravenously every 3 weeks, with an initial higher dose of 150 μg/kg followed by a reduced dose of 75 μg/kg for up to 8 cycles, distinguishing it from other treatments by its specific targeting mechanism and dosage regimen tailored to this patient population.

SUMMARY:
The goal of this clinical trial is to evaluate whether the drug Loncastuximab Tesirine can treat patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) or High-Grade B-Cell Lymphoma (HGBCL) who have not responded to or have had a relapse after CAR-T therapy. The main question it aims to answer is:

* Can Loncastuximab Tesirine improve the overall response rate (ORR) in patients who have failed CAR-T therapy?
* What are the safety and potential side effects of Loncastuximab Tesirine in this patient group?

This is a single-arm clinical trial, meaning all participants will receive the same treatment and there will be no comparison group. Researchers will focus on evaluating the effectiveness of the drug in helping patients achieve a response to treatment, and they will also assess the safety of the treatment.

Participants will:

* Be treated with Loncastuximab Tesirine through an intravenous (IV) infusion every 3 weeks for up to 8 cycles.
* Undergo regular assessments to monitor the response to treatment, including PET-CT scans and blood tests to check for markers of the disease.
* Be asked to provide informed consent before beginning the study and agree to follow the study procedures, including having biopsies performed to analyze biomarkers before starting treatment.
* Be followed for up to 2 years after completing the treatment to track their progress and response.

This study aims to help doctors understand if Loncastuximab Tesirine can offer a new treatment option for patients who have not responded to CAR-T therapy and have limited options for further treatment. The trial will also provide more information on how to manage the safety of this treatment for these patients.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the feasibility, safety, and efficacy of Loncastuximab Tesirine in patients with relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL) or High-Grade B-Cell Lymphoma (HGBCL) who have not responded to or have had a relapse following treatment with CAR-T therapy. This trial aims to assess whether Loncastuximab Tesirine can provide a viable therapeutic option for this patient population, particularly considering the urgent unmet medical need for new treatment options in cases where CAR-T therapy has failed.

Study Design: This study is a Phase II, multicenter, single-arm, prospective clinical trial. It will enroll a total of 50 patients diagnosed with DLBCL or HGBCL, who have experienced relapse or refractoriness after CAR-T therapy. The trial will focus on assessing the overall response rate (ORR), as well as the safety profile of the drug in this population.

Treatment Protocol: Loncastuximab Tesirine (also known as an antibody-drug conjugate or ADC) will be administered intravenously (IV) every three weeks for a total of up to 8 cycles, following the following dosing schedule:

150 μg/kg for the first two cycles (C1D1 and C2D1), 75 μg/kg starting from cycle 3 (C3D1) until the completion of the treatment. The drug will be infused over a 30-minute period. Patients will be closely monitored for adverse events during each infusion, and the dosage will be adjusted as needed based on safety and tolerability.

Study Objectives: The primary objective of this clinical trial is to evaluate the efficacy of Loncastuximab Tesirine in patients with relapsed or refractory DLBCL or HGBCL who have not responded to CAR-T therapy, as measured by the overall response rate (ORR). The secondary objectives of the study are to assess progression-free survival (PFS), overall survival (OS), and duration of response (DOR). Additionally, the trial will focus on the safety and tolerability of the drug, as well as exploring the relationship between biomarkers and clinical outcomes.

The primary hypotheses to be tested in this trial are:

The ORR for patients treated with Loncastuximab Tesirine is greater than 30%, with a goal of reaching 45%.

The treatment will be well-tolerated, with manageable side effects in this patient population.

The study will also investigate exploratory objectives, including the assessment of changes in disease markers (e.g., LDH, CRP, ferritin) and their correlation with clinical outcomes, as well as exploring changes in circulating tumor DNA (ctDNA) as a potential biomarker of treatment response.

Eligibility and Enrollment: Eligible participants will be adults aged 18 years or older who have been diagnosed with relapsed or refractory DLBCL or HGBCL, and who have not responded to or have relapsed after CAR-T therapy. Detailed criteria for inclusion and exclusion are outlined in the study's protocol, which focuses on ensuring that participants are in an appropriate health condition to receive the treatment and can be closely monitored for the duration of the study.

Informed Consent and Screening: Before beginning the treatment, all participants must provide written informed consent. Screening will involve a series of assessments, including a review of the patient's medical history, laboratory tests, imaging studies (such as PET-CT or CT scans), and biomarker analysis to ensure they meet the eligibility criteria.

In particular, a biopsy of the tumor tissue will be required before enrollment for biomarker analysis, and tests such as a negative pregnancy test will be mandatory for women of childbearing age. Participants will also need to have adequate organ function and a performance status (ECOG) between 0 and 2.

Study Procedures:

Initial Assessment (Screening): Participants will undergo a screening period during which baseline assessments are conducted. This includes a full medical history review, laboratory tests (such as blood counts, liver and kidney function tests), imaging studies (such as PET-CT scans), and the collection of tumor tissue samples for biomarker analysis.

Treatment Cycle: The treatment will involve administration of Loncastuximab Tesirine via intravenous infusion every 21 days (three-week intervals) for up to 8 cycles. Each infusion will be monitored for potential allergic reactions and adverse effects. Patients will be closely observed for 30 minutes following the infusion, and any adverse reactions will be managed as appropriate. Patients will also have regular clinical evaluations, including blood work, to monitor for treatment-related toxicities.

Response Evaluation: The effectiveness of the treatment will be evaluated based on changes in the size of the tumor as determined by imaging studies (PET-CT or CT scans). This will be performed at various timepoints: after Cycle 1 Day 1 (C1D1), before Cycle 3 Day 1 (C3D1), and at the end of treatment (EOT). Tumor response will be categorized as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) according to the Lugano Classification (2014).

Post-Treatment Follow-Up: After completing the treatment cycles, patients will be followed up for 2 years. Follow-up visits will include imaging (PET-CT or CT scans) and laboratory tests to monitor disease progression, as well as assessment of any long-term treatment-related side effects.

Safety Monitoring: The safety of the treatment will be closely monitored throughout the study. Vital signs, physical exams, and performance status (ECOG PS) will be assessed regularly. Blood tests will be conducted to monitor organ function (liver, kidney) and the hematologic profile (complete blood count, liver enzymes, renal function markers). The occurrence of adverse events (AE) and serious adverse events (SAE) will be recorded, and the severity of AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0).

Statistical Analysis: The study is designed to assess the efficacy of Loncastuximab Tesirine in this specific population. The sample size of 50 patients was chosen to provide sufficient statistical power to detect a significant response rate. The primary endpoint, the overall response rate (ORR), will be calculated as the proportion of patients who achieve a complete or partial response. A target ORR of 45% is considered clinically relevant, while an ORR below 30% would suggest that the treatment is not effective.

The secondary endpoints, including progression-free survival (PFS), overall survival (OS), and duration of response (DOR), will be analyzed using the Kaplan-Meier method. Differences between subgroups will be assessed using the log-rank test, and Cox regression analysis will be performed to estimate hazard ratios for survival outcomes.

The safety data will be summarized descriptively, including the frequency and severity of adverse events. The frequency of adverse events will be compared between different subgroups to identify potential risk factors for toxicity.

Exploratory Analyses: The exploratory objectives of the study include evaluating biomarkers that may help predict treatment response, such as changes in serum markers (LDH, CRP, ferritin) and the analysis of circulating tumor DNA (ctDNA). These exploratory analyses will help establish potential biomarkers for monitoring treatment response and could guide future studies on the mechanism of action of Loncastuximab Tesirine in patients with relapsed/refractory DLBCL or HGBCL.

Expected Outcomes: The study is expected to provide valuable information on the efficacy and safety of Loncastuximab Tesirine in patients with relapsed or refractory DLBCL or HGBCL who have failed CAR-T therapy. If the treatment demonstrates a significant response rate and manageable safety profile, it could potentially become a new therapeutic option for this challenging patient population.

Furthermore, the exploratory analyses of biomarkers and ctDNA will offer insights into the molecular mechanisms behind treatment response and resistance, which could be crucial for the development of personalized treatment strategies in the future.

Study Timeline:

Study Initiation: Approximately 1 month after approval by the Ethics Committee. Enrollment Period: Expected to last for 18 months, with the first patient expected to begin treatment shortly after Ethics Committee approval.

Follow-Up Period: Patients will be followed for up to 2 years after the completion of the last treatment cycle.

Data Analysis: Data analysis is expected to be completed within 3 months following the last patient's final visit, and the final study report will be available within 10-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years.
2. Ability to provide written informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Histologically confirmed diagnosis of one of the following:

   * Diffuse large B-cell lymphoma (DLBCL), non-Hodgkin lymphoma, or high grade B-cell lymphoma (HGBCL), including double/triple-hit lymphomas with MYC, BCL2, and/or BCL6 rearrangements.
   * Relapsed/refractory disease after prior CAR-T therapy, defined as:

   Progressive disease (PD) at any time following CAR-T infusion. Partial response (PR) or stable disease (SD) at 3 months post-CAR-T infusion.
5. Measurable disease as defined by the Lugano 2014 Classification and confirmed by PET-CT, CT, or MRI scans, as appropriate.
6. Previous treatment with Loncastuximab Tesirina is allowed if the patient was in complete response (CR) or partial response (PR) at the time of discontinuation of the drug.
7. Negative pregnancy test (β-HCG) for women of childbearing potential, performed within 7 days before the first dose of study drug (C1D1).
8. Female patients of childbearing potential must agree to use highly effective contraception from the time of informed consent until at least 9 months after the last dose of Loncastuximab Tesirina. Male patients with female partners of childbearing potential must agree to use highly effective contraception from the time of informed consent until at least 6 months after the last dose of Loncastuximab Tesirina.
9. Adequate renal, hepatic, pulmonary, and cardiac function:

   Creatinine clearance ≥40 mL/min. ALT/AST ≤2.5 x ULN. Total bilirubin ≤1.5 x ULN (except for patients with Gilbert's syndrome). LVEF ≥50% (or center-specific lower limit). Oxygen saturation >92% at rest and no dyspnea >Grade 1.
10. Adequate hematologic function:

Absolute neutrophil count ≥1.0 × 10⁹/L. Hemoglobin ≥9.0 g/dL. Platelets ≥50 × 10⁹/L.

Exclusion Criteria:

1. Known hypersensitivity to Loncastuximab Tesirina or any component of the drug.
2. Pregnant or breastfeeding women.
3. Active second primary malignancy, except for skin cancer, non-metastatic prostate cancer, cervical carcinoma in situ, ductal or lobular carcinoma in situ of the breast, or other malignancies that are considered not to interfere with the study by the investigator.
4. Active central nervous system (CNS) involvement, including leptomeningeal disease.
5. Tumor mass with a diameter >10 cm.
6. Positive for HIV, hepatitis B (HBV), or hepatitis C (HCV) requiring antiviral treatment.
7. Clinically significant third-space fluid accumulation (e.g., ascites or pleural effusion requiring drainage or associated with respiratory distress).
8. Significant comorbid conditions, including uncontrolled hypertension (BP ≥160/100 mmHg), unstable angina, congestive heart failure (NYHA class III or IV), recent myocardial infarction or angioplasty within 6 months prior to screening, uncontrolled arrhythmia, poorly controlled diabetes, or severe chronic lung disease.
9. Active autoimmune disease, motor neuropathy of autoimmune origin, or other autoimmune diseases affecting the central nervous system (CNS).
10. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
11. Recent chemotherapy, radiotherapy, or other anticancer treatments (within 14 days prior to study drug administration, except if approved by the Sponsor).
12. Planned administration of a live vaccine after the first dose of study drug (C1D1).
13. Use of any experimental drug or therapy within 14 days before the first dose of study drug (C1D1).
14. Failure to recover from prior chemotherapy or radiation-related toxicities to ≤Grade 1 (CTCAE v5.0) before screening.
15. Any other disease, anomaly, or medical condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study or pose a risk to the patient.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) in Patients with Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) or High-Grade B-Cell Lymphoma (HGBCL) Following Failure of CAR-T Therapy After Treatment with Loncastuximab Tesirine | The Overall Response Rate will be assessed at three key time points: 6 weeks after C1D1 (each cycle is 28 days), before C3D1, and at the end of treatment an average of 6 months. These assessments will evaluate the best OR to Loncastuximab Tesirine.
  The primary outcome measure, Overall Response Rate (ORR), is defined as the proportion of patients who achieve either a Complete Response (CR) or Partial Response (PR) to treatment with Loncastuximab Tesirine, as assessed by independent central review using the 2014 Lugano Classification criteria. CR is defined as the complete disappearance of all measurable disease, while PR indicates a significant reduction in tumor size. ORR is evaluated at several time points: 6 weeks after Cycle 1 Day 1 (each cycle is 28 days), before Cycle 3 Day 1 (C3D1), and until study treatment completion, an average of 6 months.

SECONDARY OUTCOMES:
Efficacy of Loncastuximab Tesirina in Relapsed/Refractory DLBCL or HGBCL Patients Post-CAR-T: Secondary Outcome Measure of Progression-Free Survival (PFS) | Progression-Free Survival (PFS) will be assessed at 6 weeks after C1D1, before C3D1, and at study treatment completion (an average of 6 months)), with subsequent follow-up every 3 months for 2 years to monitor disease progression or death.
  Progression-Free Survival (PFS): PFS is defined as the time from the first administration of the study drug to the first documented progression of disease (based on central review) or death from any cause. It is used to evaluate the duration of time patients remain free from disease progression while receiving treatment with loncastuximab tesirina. The metric is essential for assessing the long-term efficacy of the treatment and provides insight into the ability of loncastuximab tesirina to control disease progression after the failure of CAR-T therapy.

OTHER OUTCOMES:
Exploratory Endpoints: Evaluation of Serum Disease and Inflammation Markers, and Correlation Between Clinical Activity and ctDNA Changes in Relapsed/Refractory DLBCL or HGBCL Patients Post-CAR-T Treatment with Loncastuximab Tesirina. CRP Levels | CRP (mg/L) will be assessed at baseline, after C1D1, before C3D1, and at the EOT (after about six months), with follow-up evaluations every 3 months during the 2-year monitoring period.
  The study will assess changes in serum CRP levels to explore their relationship with clinical activity, as measured by ORR. The correlation between CRP levels and clinical activity will be explored.
Exploratory Endpoints: Evaluation of Serum Disease and Inflammation Markers, and Correlation Between Clinical Activity and ctDNA Changes in Relapsed/Refractory DLBCL or HGBCL Patients Post-CAR-T Treatment with Loncastuximab Tesirina. LDH Levels. | LDH (U/L ) will be assessed at baseline, after C1D1, before Cycle C3D1, and at the EOT( after about six months), with follow-up evaluations every 3 months during the 2-year monitoring period.
  The study will assess changes in serum LDH levels to explore their relationship with clinical activity, as measured by Objective Response Rate (ORR). The correlation between LDH levels and clinical activity will be explored.
Exploratory Endpoints: Evaluation of Serum Disease and Inflammation Markers, and Correlation Between Clinical Activity and ctDNA Changes in Relapsed/Refractory DLBCL or HGBCL Patients Post-CAR-T Treatment with Loncastuximab Tesirina. Ferritin Levels. | Ferritin (ng/mL) will be assessed at baseline, after C1D1, before C3D1, and at the EOT (after about six months), with follow-up evaluations every 3 months during the 2-year monitoring period.
  The study will assess changes in serum ferritin levels to explore their relationship with clinical activity, as measured by ORR. The correlation between ferritin levels and clinical activity will be explored.
Exploratory Endpoints: Evaluation of Serum Disease and Inflammation Markers, and Correlation Between Clinical Activity and ctDNA Changes in Relapsed/Refractory DLBCL or HGBCL Patients Post-CAR-T Treatment with Loncastuximab Tesirina. ctDNA Levels | ctDNA will be assessed at baseline, after C1D1, before C3D1, and at the EOT ( after about six months) , with follow-up evaluations every 3 months during the 2-year monitoring period.
  The study will assess changes in ctDNA levels to explore their relationship with clinical activity, as measured by ORR. The correlation between ctDNA levels and clinical activity will be explored. Units of Measure: ng/mL or copies per mL (depending on the assay used).

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria, ALESSANDRIA
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, BO
  - Azienda Sanitaria Ospedaliera Santa Croce e Carle di Cuneo, Cuneo, Cuneo
  - Ospedale San Raffaele, Milan, MILANO
  - Istituto Nazionale dei Tumori, Milan, MILANO
  - Irccs Istituto Clinico Humanitas, Rozzano, MILANO
  - AOU Policlinico Umberto I, Roma, RO

IPD SHARING:
Plan to Share IPD: No